CLINICAL TRIAL: NCT00032396
Title: A Study to Evaluate Retisert in the Treatment of Patients With the "Wet" Form of Age-Related Macular Degeneration
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Control Delivery Systems (Industry)
Collaborators: Bausch & Lomb Incorporated (Industry)
Purpose: Treatment
Other Study IDs: CDS FL-004
Record Dates: First submitted 2002-03-20; First posted 2002-03-22 (Estimated); Last update posted 2006-05-29 (Estimated); Status verified 2002-12

CONDITIONS: Macular Degeneration
Keywords: AMD; ARMD; Age-Related Macular Degeneration; Subfoveal Choroidal Neovascularization; CNV
MeSH Terms: conditions — Macular Degeneration | interventions — Fluocinolone Acetonide

INTERVENTIONS:
Drug: Retisert Implant

SUMMARY:
A study evaluating Retisert in patients with age-related macular degeneration

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-11

CONTACTS AND LOCATIONS:
Locations (1):
- Control Delivery Systems, Inc., Watertown, Massachusetts, United States